CLINICAL TRIAL: NCT06796270
Title: Efficacy and Safety of Hypofractionated Radiotherapy for Nasopharyngeal Carcinoma
Brief Title: Hypofractionated Radiotherapy for Nasopharyngeal Carcinoma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Second Affiliated Hospital of Hainan Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-K52-01
Record Dates: First submitted 2025-01-14; First posted 2025-01-28 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Nasopharyngeal Carcinoma (NPC)
Keywords: Nasopharyngeal Carcinoma (NPC); Hypofractionated radiotherapy
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — Radiation Dose Hypofractionation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hypofractionated radiotherapy (Experimental): The patients with nasopharyngeal carcinoma were given the dose of large segmentation radiotherapy, 2.64Gy/ time, 5 times/week, a total of 25 times, a total of 66Gy/5 weeks.
  Interventions: Radiation: Hypofractionated radiotherapy

INTERVENTIONS:
Radiation: Hypofractionated radiotherapy — The patients with nasopharyngeal carcinoma were given the dose of large segmentation radiotherapy, 2.64Gy/ time, 5 times/week, a total of 25 times, a total of 66Gy/5 weeks.

SUMMARY:
The purpose of this study was to evaluate the efficacy and safety of large fractionation radiotherapy in nasopharyngeal carcinoma patients, and to analyze whether Hypofractionated radiotherapy is not inferior to conventional radiotherapy.

DETAILED DESCRIPTION:
Nasopharyngeal carcinoma (NPC) is a type of head and neck malignancies with uneven geographic distribution. According to the World Health Organization, about 40 percent of nasopharyngeal cancer cases occur in China, especially in southern China. Because of the anatomical location, pathological type and biological behavior of nasopharyngeal carcinoma, radiotherapy is the most important treatment method for nasopharyngeal carcinoma. There are four main factors that affect the effect of radiotherapy: (1) repair of radiation damage, (2) repopulation or reproliferation of tumor cells, (3) reoxygenation of hypoxic tumor cells, and (4) redistribution of cell cycle. Reproliferation of surviving tumor cells is one of the important reasons for local failure of conventional frit radiotherapy. The key to improve local control of tumor cells is to overcome the accelerated reproliferation of tumor cells.

Under the conditions of conventional radiotherapy techniques, the organs can be exposed to a large range of radiation, serious damage, difficult to achieve the target dose, and lead to some acute and late toxicity, which may have a negative impact on the patient's quality-of-life (QoL). The conventional segmentation course is too long and the treatment time is too long, thus creating conditions for the accelerated reproliferation of tumor cells, which is not conducive to local control, and has a certain impact on patients in physiological, psychological and economic aspects.

Clinical studies have shown that a variety of human tumors have accelerated reproliferation after conventional radiotherapy, and this reproliferation is closely related to the potential doubling time of tumors. Hypofractionated radiotherapy , also known as low segmentation radiotherapy, refers to the dose segmentation mode with a single radiotherapy dose >2Gy. It can shorten radiotherapy on the premise that the biological effect dose of conventional dose segmentation radiotherapy is equivalent to or increased. It has been widely used in the treatment of a variety of tumors, and is a safe, effective and short course of radiotherapy mode. This method can increase the single dose and shorten the course of treatment, considering the reproliferation of tumor cells and the protection of normal tissues, which is in line with the principle of radiobiology. When the time factor of doubling time days was added, the large segmentation radiotherapy was higher than that of conventional radiotherapy and was consistent with clinical results. Recently, many scholars have made clinical exploration on the technique of Hypofractionated radiotherapy, which provides a new model for radiotherapy. Compared with conventional segmentation, Hypofractionated radiotherapy can give a higher bioeffective dose to the tumor, effectively improve the tumor control rate, shorten the average radiotherapy time by one week, and reduce the reproliferation of tumor cells.

In recent years, with the increasingly detailed optimization of precision radiotherapy technology and the development of radiobiology, Hypofractionated radiotherapy has achieved good therapeutic effects in prostate cancer, lung cancer, liver cancer and breast cancer. Long Bin et al. found that in patients with recurrent nasopharyngeal carcinoma, the duration of Hypofractionated radiotherapy is significantly shorter than that of conventional fractionated radiotherapy, which reduces part of the radiation damage reaction, increases the equivalent biological dose, and can significantly increase the Tumor Control Probability (TCP), with good short-term and long-term efficacy. High gain ratio and good safety were obtained. At present, there is no research on Hypofractionated radiotherapy in nasopharyngeal carcinoma patients at home and abroad. At present, conventional segmentation is still advocated, and the conventional mode is 70Gy/35F/7W. However, this dose segmentation mode has negative factors such as multiple patient trips and high medical costs. Radiobiology and a large number of clinical studies have shown that there is accelerated proliferation of tumor cells after radiotherapy, and this accelerated reproliferation is the main reason for radiotherapy failure, thus challenging whether conventional fractionated radiotherapy is the best scheme. A variety of unconventional fractionated radiotherapy schemes such as hyperfractionation, Hypofractionated radiotherapy and late accelerated fractionation have been proposed to improve the therapeutic effect of cancer.

Therefore, we initiated a non-inferior, non-randomized controlled clinical trial to evaluate whether mafrit is comparable to conventional radiotherapy in nasopharyngeal carcinoma patients with a view to further improving the prognosis and quality of life of nasopharyngeal carcinoma patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 years, male or female；
2. Performance status ≤ 2 ;
3. Nasopharyngeal cancer patients diagnosed by pathology (including histology or cytology) , of nasopharyngeal non-keratonic carcinoma (differentiated or undifferentiated, whether TNM staging);
4. Have at least one evaluable lesion (according to Recist1.1 criteria)
5. Expected survival ≥6 months.
6. The main organs are functioning normally and meet the following standards: (1) Blood routine examination must meet the following criteria: (no blood transfusion within 14 days) a. HB ≥ 100g/L, b. WBC ≥3×10^9/L c. ANC≥1.5×10^9/L, d. PLT ≥100×10^9/L; (2) Biochemical examination must meet the following standards: a. BIL<1.5 times the upper limit of normal value (ULN), b. ALT and AST<2.5ULN, GPT ≤1.5×ULN; c. Serum Cr≤1 ULN, endogenous creatinine clearance rate>60ml/min (Cockcroft Gault formula);(3).Good coagulation function: defined as International standardized ratio (INR) or prothrombin time (PT) ≤1.5×ULN;(4).The myocardial enzyme spectra were in the normal range.
7. Patients willing and able to give signed informed consent and, in the opinion of the Investigator, to comply with the Clinical Investigation Plan tests and procedures.

Exclusion Criteria:

1. Pregnant or lactating women
2. As determined by the investigators, there were severe comorbidities that could not tolerate or complete radiation therapy.
3. There are contraindications in MRI;
4. Second primary malignancy exists;
5. Patients with severe complications,such as hypertension, coronary heart disease,mental disease or patients who had any allergies before;
6. Received any other research in the past 4 weeks before enrollment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2026-02-20 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | 3 months， 6 months，12 months，24 months，36 months，60 months
  overall response rate (ORR) in patients with nasopharyngeal carcinoma treated with Hypofractionated radiotherapy

SECONDARY OUTCOMES:
Overall survival (months) | 3 months， 6 months，12 months，24 months，36 months，60 months
  This is defined as the number of months participants survived from completion date of radiation therapy until the date of death. If a participant is alive, the participant censored at the date of last documentation of the patient being alive.
Progress-free survival (months) | 3 months， 6 months，12 months，24 months，36 months，60 months
  This is defined as the number of months participants experienced no locoregional recurrence or distant metastasis from completion date of radiation therapy until the date of progression. The date of progression will be defined as the date of initial suspicion for progression by physical exam or imaging studies.Evaluation of Incidence of Treatment-Emergent Adverse Events Patients will be educated and instructed to report any adverse events
Number acute toxicities | 1-2 weeks, 3 months, 6 months
  Number of acute toxicities associated with radiation experienced by participants based on the follow-up assessments at 1-2 weeks, 3 months, 6 months following radiation therapy completion
Number of chronic toxicities | 2 weeks, 3 months, 6 months and 12 months
  Number of chronic toxicities associated with radiation experienced by participants based on the follow-up assessments completed at 2 weeks, 3 months, 6 months and 12 months following radiation therapy
Patient reported Health related quality of life (HRQoL) | 2 months
  Patient reported health related quality of life is captured through a questionnaire the Generic European Organization for Research and Treatment of Cancer (EORTC) QLQ-C30. It is a core scale applicable to all cancer patients. It contains a total of 30 items, items 1 to 28 are divided into 4 grades and scored 1 to 4 points, items 29 and 30 are divided into 7 grades and scored 1 to 7 points. The 30 entries are divided into 15 domains, including 5 functional domains (i.e., somatic, role, cognitive, emotional, and social), 3 symptom domains (i.e., fatigue, pain, nausea, and vomiting), 1 quality of life domain, and 6 single entries/domains. A high score on functional or global health status scale represents a high/healthy level of functioning
Tolerance and compliance | 2 months
  The number of patients who received the full course of Hypofractionated radiotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: yuecan zeng, doctor, Study Director — The Second Affiliated Hospital of Hainan Medical University
Locations (1):
- The Second Affiliated Hospital of Hainan Medical University, Haikou, Hainan, China